CLINICAL TRIAL: NCT00506337
Title: Evaluation of Effect of Integrated Treatment by Traditional Chinese and Western Medicine for Severe Acute Pancreatitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Collaborators: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006BAI04A15
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Pancreatitis, Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Qingyi granules — Control group: The therapeutic methods accord to the concert schemes cited in the "Guides to diagnosis and treatment of severe acute pancreatitis" introduced by the Pancreatic Surgery Group of Surgical Chapter of Chinese Medical Association.
  Treatment group: In addition to the concert schemes cited in the "Guides to diagnosis and treatment of severe acute pancreatitis", during the first stage of the disease herbal Qingyi granules 1-B 4 bags dissolved in water 200ml were administered through the gastric tube q6h. Then the gastric tube was closed for 1h, and Qingyi granules 1-B another 4 bags dissolved in water 400ml were given through enema q6h. During the second stage (from the 2nd week to the 4th week after onset) Qingyi granules 2-B 2bags dissolved in water 200ml were added QD.

SUMMARY:
With multicenter randomized control clinical evaluation investigations, the scheme of integrated medicine treatment of severe acute pancreatitis (SAP) was further improved, and the therapeutic effects, safety and indications assured. Drawing in latest research fruits at home and abroad, a clinical practical guideline for integrated medicine of diagnosis and treatment of SAP would be formed, to be popularized all over China.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18yr-70yr, complying with the diagnostic standard of acute pancretitis (clinical symptoms and signs, elevated blood and urine amylase, and imaging criteria), conforming to 3 or more Ranson's criteria and APACHE-II score larger than 8, Balhazar CT score larger than 5.

Exclusion Criteria:

* Pregnancy, nursing mother, critical cases of advanced tumor, on the verge of death (estimated to be moral in 12h), severe visceral function disturbance, patients undergoing other therapeutic research that might interfere with the present study.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-10; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
1,Mortality 2,Morbidity 3,Crossing stage cure rates 4,Number of operation procedures 5,Incidences of secondary infections 6,Hospitalization days 7,Total expenses 8,Traditional Chinese medicine diagnostic parameters | To observe the relationship between the parameters of the first and second stages and the endpoints

SECONDARY OUTCOMES:
1.Routine laboratory tests, blood and urine amylase, blood lipase. 2.Important visceral function criteria 3.microorganism culture, endotoxin determination, CRP 4.B-ultrasound, CT, chest films, plain abdomen film | The above criteria should be tested on admission, and 24h, 48h and 72h later, 5d, 7d, and 2wks after admission, and on the day of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Naiqiang Cui, Dr, Principal Investigator — Tianjin Nankai Hospital; Qing Xia, Dr, Principal Investigator — West China Hospital; Qinghui Qi, Dr, Principal Investigator — The 1st Affiliated Hospital, Dalian Medical Unversity
Locations (3):
- China (3):
  - The 1st Affiliated Hospital, Dalian Medical Unversity, Dalian, Liaoning
  - West China Hospital, Sichuan Unversity, Chengdu, Sichuan
  - Tianjin Nankai Hospital, Tianjin